CLINICAL TRIAL: NCT04267900
Title: 99mTc-HPArk2 SPECT/CT for the Detection of HER2-positive Breast Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PekingUMCH-NM25
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Breast Cancer
Keywords: SPECT/CT; HER2 imaging
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 99mTc-HPArk2 SPECT/CT (Experimental): The patients were injected with 11.1 (MBq) per kilogram body weight of 99mTc-HPArk2 in one dose intravenously and underwent SPECT/CT scan 30-60 min later.
  Interventions: Drug: 99mTc-HPArk2

INTERVENTIONS:
Drug: 99mTc-HPArk2 — 99mTc-HPArk2 were injected into the patients before the SPECT/CT scans
  Other Names: 99mTc labelled HER2 affibody

SUMMARY:
This is an open-label single photon emission tomography/computed tomography (SPECT/CT) study to investigate the diagnostic performance and evaluation efficacy of 99mTc-HPArk2 in breast cancer patients. A single dose of 11.1Mega-Becquerel (MBq) per kilogram body weight 99mTc-HPArk2 will be injected intravenously. Visual and semiquantitative method will be used to assess the SPECT/CT images.

DETAILED DESCRIPTION:
99mTc-HPArk2 is an affibody probe targeting HER2. The investigators will determine the use of 99mTc-HPArk2 SPECT/CT in the detection of HER2-positive breast cancer, and to compare its diagnostic value with routine immunohistochemistry (IHC) pathological staining. HER2 imaging, specifically to HER2 receptor expressed on malignant breast cancer cell surface, might help for targeted therapy with monoclonal antibody such as trastuzumab in breast cancer, and may improve the treatment strategy of breast cancer. The investigator will determine the use of 99mTc-HPArk2 SPECT/CT in stratifying breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* patients in suspicion of breast cancer by mammography or ultrasonography,and being able to provide basic information and sign the written informed consent form

Exclusion Criteria:

* The exclusion criteria included claustrophobia, pregnancy, breastfeeding, kidney or liver failure, inability to fulfill the study, and undergoing any preceding local or systemic therapies that might interfere with HER2 binding.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-12-07 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Standardized uptake value of 99mTc-HPArk2 in breast tumor | 1 year
  The semiquantitative analysis will be performed by the same person for all the cases, and the standardized uptake value (SUV) of the tracer in breast tumor will be measured. SUV were obtained by a self-made software and referring to phantom study.

SECONDARY OUTCOMES:
Adverse events collection | 1 week
  Adverse events within 1 week after the injection and scanning of patients and patients will be followed and assessed

CONTACTS AND LOCATIONS:
Overall Officials: Zhaohui Zhu, MD,PHD, Study Chair — Peking Union Medical College Hospital, Chinese Academy of Medical Science and Peking Union Medical College
Locations (1):
- Peking Union Medical College Hospital, Chinese Academy of Medical Science and Peking Union Medical College, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Shi J, Du S, Wang R, Gao H, Luo Q, Hou G, Zhou Y, Zhu Z, Wang F. Molecular imaging of HER2 expression in breast cancer patients using a novel peptide-based tracer 99mTc-HP-Ark2: a pilot study. J Transl Med. 2023 Jan 11;21(1):19. doi: 10.1186/s12967-022-03865-y. PMID 36631812